CLINICAL TRIAL: NCT05718154
Title: Comparison Between the Incidence of Assault-induced Trauma in Patients Attending to Trauma Unit in Assiut University Hospital and Trauma Unit in Suez Canal University Hospital
Brief Title: Comparing the Incidence of Assault-Induced Trauma Patients in Assiut University and Suez Canal University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abdelzaher, principal investigator, Assiut University
Other Study IDs: AIT in Assiut and Suez Canal
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-02

CONDITIONS: Assault

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assault-Induced Trauma Patients in Suez Canal University Hospital-Trauma Unit: Total coverage of all patients fulfilled the inclusion criteria
  * From April 2023 to September 2023 in Suez Canal University Hospital, Emergency Department.
- Assault-Induced Trauma Patients in Assiut University Hospital-Trauma Unit: Total coverage of all patients fulfilled the inclusion criteria
  * From October 2023 to March 2024 in Assiut University Hospital, Trauma Unit.

SUMMARY:
Aim of this research is to compare between the incidence of assault-induced trauma in patients attending to trauma unit at Assiut University Hospital and trauma unit at Suez Canal University Hospital

DETAILED DESCRIPTION:
Trauma is the third leading cause of death in all age groups after cardiovascular diseases and cancer. However, trauma is the most common cause of death in the age of first four decades. There are many types of major trauma, an important one of which is the assault-induced trauma.

Assault-Induced Trauma is a potentially life-threatening emergency that often requires a multidisciplinary approach, as Assault-Induced Trauma can contribute substantially to death, permanent disability and chronic illness.

Assault may be said to be intentional violent bodily contact with another person without consent. Assault occurs when an individual or a group provokes and attacks another person with or without the use of a weapon.

Injuries yield from such type of trauma are variable and complex, with the predominance of young males as a victims. Wide variety of injuries range from isolated wound to complex injuries affecting multi-organs.

According to the severity of Assault-Induced injuries and the need for more diagnostic and therapeutic intervention hospital stay can be determined for those patients.

Studies conducted in the USA for analysis of non-fatal assault injuries has shown that 87% of patients were treated and discharged without the need for inpatient admission.

With the improvement in the approach adopted for treatment of assaulted patients, treatment modalities have shifted toward a more conservative approach than an invasive approach that was practiced previously.

Assault induced injuries commonly caused by the use of body force, blunt trauma and sharp objects.

Previous studies done has shown that male gender in their 20s and 30s is a high risk groups and showed also that incidence is related to the economic and political state of the community.

Studies done in Europe and United Kingdom demonstrated that factors such as unemployment, low socioeconomic status and alcohol consumption increase assault rates. On the other hand, high level of education serves as a positive protective factor against Assault prevalence.

Late reports in USA demonstrates the decline in nonfatal assault injuries among young population compared to previous analyses.

The decline refers to increased implementation and beneficial outcome of evidence-based prevention strategies that reach young patients in USA.

Unfortunately, there is no previous studies in our community discussing this problem and there is no recent official statistics that can help in determining how huge the problem is, and point to the factors that can be taken as a base to the future plans to solve the problem.

This study aims to characterize cases of assault-induced trauma victims presenting to trauma unit in Assiut University Hospital in comparison to trauma unit in Suez Canal University Hospital. This will aid in analysis of the incidence of the problem and estimate the effectiveness of current management methods.

Presence of such type of researches will enhance the health service delivered to targeted groups and will encourage further researches.

ELIGIBILITY:
Inclusion Criteria:

Assault-induced trauma cases admitted to the emergency unit and ICU department of:

* All age groups.
* During one year from the start of the study(6 months in Suez Canal University Hospital and 6 months in Assiut University Hospital).
* Victims with isolated wound or complex injuries

Exclusion Criteria:

* Self-inflicted injuries.
* Accidental injuries.
* Patients with insufficient data.
* Victims of assault who died prior to their arrival at the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total coverage of all patients fulfilled the inclusion criteria
  * From April 2023 to September 2023 in Suez Canal University Hospital, Emergency Department.
  * From October 2023 to March 2024 in Assiut University Hospital, Trauma Unit.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Comparing the incidence of cases in number(N) | a year from the start of the study
  Compare between the incidence of assault-induced trauma in patients attending to trauma unit in Assiut University Hospital and Suez Canal University Hospital in number(N).

SECONDARY OUTCOMES:
Describing demographics, mode and management | a year from the start of the study
  Describing demographics(Age(number of cases in each age group and mean age of incidence), Gender(number of male and female cases(n) and its percentage(%)), Nationality(number of Egyptian and non Non-Egyptian cases(n)and its percentage) ), mode(bodily force, sharp object, blunt object, gun shoot, explosives, unknown in number(n) and Percentage(%) )and management(surgical, procedural, conservative cases in number(n) and percentage(%) )of assault-induced trauma in order to be used as a base for future plans to decrease the incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hani Elmorabaa, Professor, Study Chair — Anesthesia and ICU department Assiut university hospital; zeinab Mohamed, Lecturer, Study Director — Emergency Medicine department, Suez Canal university, Ismailia

REFERENCES:
- [Background] Olojede A, Gbotolorun OM, Ogundana OM, Emeka IC, Emmanuel MM, Oluseye S, Runsewe O. PATTERN OF ASSAULT-RELATED MAXILLOFACIAL INJURIES TREATED AT THE GENERAL HOSPITAL, LAGOS, NIGERIA. J West Afr Coll Surg. 2016 Jul-Sep;6(3):68-82. PMID 28856125
- [Background] Kristoffersen S, Normann SA, Morild I, Lilleng PK, Heltne JK. The hazard of sharp force injuries: Factors influencing outcome. J Forensic Leg Med. 2016 Jan;37:71-7. doi: 10.1016/j.jflm.2015.10.005. Epub 2015 Nov 5. PMID 26599374
- [Background] Tingne CV, Shrigiriwar MB, Ghormade PS, Kumar NB. Quantitative analysis of injury characteristics in victims of interpersonal violence: an emergency department perspective. J Forensic Leg Med. 2014 Aug;26:19-23. doi: 10.1016/j.jflm.2014.06.003. Epub 2014 Jun 11. PMID 25066168
- [Background] David-Ferdon CF, Haileyesus T, Liu Y, Simon TR, Kresnow MJ. Nonfatal Assaults Among Persons Aged 10-24 Years - United States, 2001-2015. MMWR Morb Mortal Wkly Rep. 2018 Feb 9;67(5):141-145. doi: 10.15585/mmwr.mm6705a1. PMID 29420463
- [Background] Bieler D, Franke AF, Hentsch S, Paffrath T, Willms A, Lefering R, Kollig EW; TraumaRegister DGU. [Gunshot and stab wounds in Germany--epidemiology and outcome: analysis from the TraumaRegister DGU(R)]. Unfallchirurg. 2014 Nov;117(11):995-1004. doi: 10.1007/s00113-014-2647-7. German. PMID 25398509
- [Background] Bass P, Sanyang E, Lin MR. Risk Factors for Violent Injuries and Their Severity Among Men in The Gambia. Am J Mens Health. 2018 Nov;12(6):2116-2127. doi: 10.1177/1557988318794524. Epub 2018 Aug 19. PMID 30124092
- [Background] Al-Busaidi M, Al-Miskry H, Al-Harbi A, Al-Zadjali I, Al-Saidi F, Al-Qadhi H. Overview of Assault-Induced Trauma Presenting to a Trauma Centre in Oman. Sultan Qaboos Univ Med J. 2021 Nov;21(4):549-553. doi: 10.18295/squmj.4.2021.033. Epub 2021 Nov 25. PMID 34888073
- [Background] Ferreira MC, Batista AM, Ferreira Fde O, Ramos-Jorge ML, Marques LS. Pattern of oral-maxillofacial trauma stemming from interpersonal physical violence and determinant factors. Dent Traumatol. 2014 Feb;30(1):15-21. doi: 10.1111/edt.12047. Epub 2013 May 15. PMID 23675634
- [Background] Faergemann C, Lauritsen JM, Brink O, Skov O, Mortensen PB. Demographic and socioeconomic risk factors of adult violent victimization from an accident and emergency department and forensic medicine perspective: a register-based case-control study. J Forensic Leg Med. 2009 Jan;16(1):11-7. doi: 10.1016/j.jflm.2008.05.014. Epub 2008 Aug 12. PMID 19061843
- [Background] Office of Juvenile Justice and Delinquency Prevention. Statistical briefing book. Washington, DC: US Department of Justice, Office of Juvenile Justice and Delinquency Prevention; 2017.
- [Background] Bell TM, Qiao N, Jenkins PC, Siedlecki CB, Fecher AM. Trends in Emergency Department Visits for Nonfatal Violence-Related Injuries Among Adolescents in the United States, 2009-2013. J Adolesc Health. 2016 May;58(5):573-5. doi: 10.1016/j.jadohealth.2015.12.016. Epub 2016 Feb 20. PMID 26907850
- [Background] David-Fredon C, Vivolo-Kantor AM, Dahlberg LL, Marshall KJ, Rainford N, Hall JE. A comprehensive technical package for the prevention of youth violence and associated risk behaviors. Atlanta, GA: US Department oh Health and Human Services, CDC; 2016.